CLINICAL TRIAL: NCT03533790
Title: DEP-ruxolitinib Regimen as a Salvage Therapy for Refractory/Relapsed Hemophagocytic Lymphohistiocytosis
Brief Title: DEP-Ru Regimen as a Salvage Therapy for HLH
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Clinical Professor, Beijing Friendship Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DEP-Ru HLH
Record Dates: First submitted 2018-05-12; First posted 2018-05-23 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Hemophagocytic Lymphohistiocytosis
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DEP-Ru (Experimental): doxorubicin (doxorubicin hydrochloride liposome injection) 25 mg/m2 day 1; etoposide 100 mg/m2 was administered day1; methylprednisolone 2 mg/kg days 1 to 5,then gradually reduce; ruxolitinib 0.3mg/kg/d。This regimen was repeated after 2 weeks.
  Interventions: Drug: DEP-Ru

INTERVENTIONS:
Drug: DEP-Ru — * Drug: ruxolitinib
  * Drug: doxorubicin
  * Drug: etoposide
  * Drug: methylprednisolone

SUMMARY:
This study aimed to investigate the efficacy and safety of ruxolitinib together with liposomal doxorubicin, etoposide and methylprednisolone (DEP-Ru) as a salvage therapy for refractory/relapsed hemophagocytic lymphohistiocytosis.

ELIGIBILITY:
Inclusion Criteria:

1. meet HLH-04 diagnostic criteria;
2. treated with HLH-94 no less than 2 weeks before enrollment and did not achieve at least PR; or relapsed patients after remission；
3. Life expectancy exceeds 1 month;
4. Age≥1 year old and ≤70 years old, gender is not limited；
5. Before the start of the study, total bilirubin ≤ 10 times the upper limit of normal; serum creatinine ≤ 1.5 times normal；
6. Serum HIV antigen or antibody negative；
7. HCV antibody is negative, or HCV antibody is positive, but HCV RNA is negative；
8. Both HBV surface antigen and HBV core antibody were negative. If any of the above is positive, peripheral blood hepatitis B virus DNA titer should be detected, and less than 1×103 copies/ml can enter the group；
9. Echocardiographic examination of LVEF ≥ 50%;
10. Informed consent.

Exclusion Criteria:

1. Heart function above grade II (NYHA)；
2. Accumulated dose of doxorubicin above 300mg/m2 or epirubicin above 450mg/m2；
3. Pregnancy or lactating Women；
4. Allergic to Pegaspargase, doxorubicin or etoposide；
5. Active bleeding of the internal organs；
6. uncontrollable infection；
7. Serious mental illness;
8. Non-melanoma skin cancer history;
9. Patients unable to comply during the trial and/or follow-up phase;
10. Participate in other clinical research at the same time.

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2018-06 (Estimated); Primary Completion 2018-06 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of treatment response | Change from before and 2,4,6 and 8 weeks after initiating DEP-Ru salvage therapy
  A complete response was defined as normalization of all of the quantifiable symptoms and laboratory markers of HLH, including levels of sCD25, ferritin, and triglyceride; hemoglobin; neutrophil counts; platelet counts; and alanine aminotransferase (ALT). A partial response was defined as at least a 25% improvement in 2 or more quantifiable symptoms and laboratory markers as follows: sCD25 response was>1.5-fold decreased; ferritin and triglyceride decreased at least 25%; for patients with an initial neutrophil count of<0.5 ×109/L, a response was defined as an increase by at least 100% to>0.5× 109/L; for patients with a neutrophil count of 0.5 to 2.0 × 109/L, an increase by at least 100% to >2.0 × 109/L was considered a response; and for patients with ALT >400 U/L, response was defined as an ALT decrease of at least 50%.

SECONDARY OUTCOMES:
Survival | from the time patients received DEP-Ru salvage therapy up to 24 months or June 2021
  survival
Adverse events that are related to treatment | through study completion, an average of 2 years
  Adverse events including myelosuppression, infection, bleeding and so on.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Background] Broglie L, Pommert L, Rao S, Thakar M, Phelan R, Margolis D, Talano J. Ruxolitinib for treatment of refractory hemophagocytic lymphohistiocytosis. Blood Adv. 2017 Aug 17;1(19):1533-1536. doi: 10.1182/bloodadvances.2017007526. eCollection 2017 Aug 22. PMID 29296794
- [Result] Wang Y, Huang W, Hu L, Cen X, Li L, Wang J, Shen J, Wei N, Wang Z. Multicenter study of combination DEP regimen as a salvage therapy for adult refractory hemophagocytic lymphohistiocytosis. Blood. 2015 Nov 5;126(19):2186-92. doi: 10.1182/blood-2015-05-644914. Epub 2015 Aug 19. PMID 26289641
- [Derived] Wang J, Zhang R, Wu X, Li F, Yang H, Liu L, Guo H, Zhang X, Mai H, Li H, Wang Z. Ruxolitinib-combined doxorubicin-etoposide-methylprednisolone regimen as a salvage therapy for refractory/relapsed haemophagocytic lymphohistiocytosis: a single-arm, multicentre, phase 2 trial. Br J Haematol. 2021 May;193(4):761-768. doi: 10.1111/bjh.17331. Epub 2021 Feb 9. PMID 33559893